CLINICAL TRIAL: NCT06891989
Title: Effects of a Mobile App-Based Mindfulness Intervention in Persons with Spinal Cord Injury and Chronic Pain: a Randomized Controlled Trial
Brief Title: Effects of a Mobile App-Based Mindfulness Intervention in Persons with Spinal Cord Injury and Chronic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Radha Korupolu, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-25-0005
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Mindfulness; Methods

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness meditation (MM) (Experimental)
  Interventions: Other: Mindfulness meditation (MM) Intervention
- Active Control (AC) (Active Comparator)
  Interventions: Other: Health Education Active Control Intervention

INTERVENTIONS:
Other: Mindfulness meditation (MM) Intervention — Participants will be asked to download the Mindfulness Coach app that provides simple instructions and brief meditation exercises.This is a a gradual training program of 14 levels which will be completed in the first 2-3 weeks. Each level provides short readings about mindfulness and one or two guided meditations (a silent "seated practice" for increasing lengths of time plus typically an additional 8-13-minute meditation). As participants progress through the levels, they earn "badges" displayed in the app, and an image of a tree on the home screen grows as each successive level is completed.For the remaining weeks of the intervention, participants will select at least one (and ideally two) guided meditation per day from the complete list of available meditations.Participants will track their progress through weekly logs.
  Arms: Mindfulness meditation (MM)
Other: Health Education Active Control Intervention — Participants will be asked to download and use the free TED Talk app, which will have 50 TED talk videos related to health that range from 3-20 minutes. Participants will be asked to watch or listen to these videos for ≥ 10 minutes daily for 6 days per week and complete weekly logs of the TED Talk app use.
  Arms: Active Control (AC)

SUMMARY:
The purpose of this study is to evaluate the efficacy of a 6-week app-guided MM intervention compared to a 6-week app-guided health education AC condition on pain intensity, pain interference, depression, and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic SCI of at least 6 months duration
* Chronic pain [defined as pain lasting at least 3 months with a pain intensity rating of 4 or higher on a 10-point visual analog scale]
* Understand spoken and written English sufficiently to provide informed consent, participate in the intervention and complete study surveys

Exclusion Criteria:

* Lack of daily internet access
* inability to demonstrate comprehension of informed consent by correctly answering 4 out of 5 questions about the study
* Significant visual/hearing impairment that does not allow use of the MM app's audiovisual presentations
* Use of any meditation more than once a week in the last 3 months
* Inability to provide or obtain an email address for registration to the AC intervention and/or communication with study staff
* inability to provide a phone number for communication with study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain intensity in people with spinal cord injury (PwSCI) as assessed by Numeric Rating Scale (NRS). | baseline , post-intervention (6 weeks after baseline)
  Pain will be measured on Numeric Rating Scale (NRS) from 0(no pain) to 10(pain as bad as you can imagine)

SECONDARY OUTCOMES:
Change in pain interference as assessed by the Spinal Cord Injury - Quality of Life (SCI-QOL) Pain Interference scale | baseline , post-intervention (6 weeks after baseline)
  This is a 10 item questionnaire, each item is typically scored on a 5-point Likert scale from 1 (Not at all) to 5 (Very much), for a maximum raw score of 50, higher scores reflect greater pain interference.
Change in depression as assessed by the Patient Health Questionnaire (PHQ-9) | baseline , post-intervention (6 weeks after baseline)
  This is a 8 item questionnaire , each measured on a 4 point scale from 0(not at all) to 3(nearly every day), for a score range of 0-27, higher score indicating worse outcome
Change in anxiety as assessed by the Generalized Anxiety Disorder (GAD-7) | baseline , post-intervention (6 weeks after baseline)
  This is an 7 item questionnaire, each is scored from 0(not at all) to 3(nearly every day), for a maximum score of 21, a higher score indicating more anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Radha Korupolu, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No